CLINICAL TRIAL: NCT02773316
Title: 2-cohort, 3-part, Open-label, Randomised, Single Dose, Crossover Study in Healthy Subjects to Compare PK & Bioavailability of a Single Dose, in Fed and Fasted State, of MR902 Prolonged Release (PR) Tablets With Immediate Release (IR) Morphine Sulfate Oral Solution
Brief Title: Study to Assess Pharmacokinetic (PK), Bioavailability & Food Effect of MR902 Compared With Immediate Release (IR) Morphine Sulphate Oral Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MR902-1501
Record Dates: First submitted 2016-05-10; First posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Opioid Substitution Treatment
MeSH Terms: interventions — Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MR902 50/0.5 mg (Experimental): MR902 50/0.5 mg PR tablets, single dose oral
  Interventions: Drug: MR902
- MR902 200/2 mg (Experimental): MR902 200/2 mg PR tablets, single dose oral
  Interventions: Drug: MR902
- IR morphine sulphate 10 mg/5mL solution (Active Comparator): IR morphine sulphate 10 mg/5mL solution, single dose oral
  Interventions: Drug: IR morphine sulphate

INTERVENTIONS:
Drug: MR902
  Arms: MR902 200/2 mg; MR902 50/0.5 mg
Drug: IR morphine sulphate
  Other Names: IR morphine sulphate 10 mg/mL solution
  Arms: IR morphine sulphate 10 mg/5mL solution

SUMMARY:
A study to assess bioavailability of a single dose of MR902 and to assess the effect of food on absorption

DETAILED DESCRIPTION:
Volunteers will receive a single dose of the investigational drug on 2 occasions and a reference drug on 1 occasion. Volunteers will be randomised to one of two groups, each group receiving a different dose strength of MR902 in fed and fasted state.

The study involves a screening visit 21 days before first dosing and 3 overnight stays in 3 study periods, and a post-study medical visit.

Volunteers will receive naltrexone to reduce anticipated opioid side effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and free of significant abnormal findings as determined by medical history, physical examination, vital signs, laboratory tests and ECG.
* Body weight ranging from 55 to 100 kg and a BMI ≥ 18.5 and ≤ 30.0.
* Willing to eat all the food supplied throughout the study.
* The subject's primary care physician has confirmed within the last 12 months of first dosing that there is nothing in their medical history that would preclude their enrolment into a clinical study.

Exclusion Criteria:

* Female subjects who are pregnant or lactating.
* Any history of drug or alcohol abuse, misuse, physical or psychological dependence.
* Any history of conditions that might interfere with drug absorption, distribution, metabolism or excretion.
* Use of opioid or opioid antagonist-containing medication in the past 30 days.
* Any history of frequent nausea or vomiting regardless of etiology.
* Any history of seizures or symptomatic head trauma.
* History of respiratory depression, hypoxia or elevated carbon dioxide levels in the blood.
* History of paralytic ileus, gastrointestinal disease or other clinically significant gastrointestinal problems.
* Participation in a clinical drug study during the 90 days preceding the initial dose in this study.
* Any significant illness during the 4 weeks preceding entry into this study.
* Use of any medication including vitamins, herbal and/or mineral supplements during the 7 days preceding the initial dose or during the course of this study (with the exception of the continued use of HRT and contraceptives).
* History of smoking within 60 days of IMP administration and refusal to abstain from smoking during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Measure the observed maximum plasma or serum concentration after administration (Cmax) | Pre-dose to 24 hours post-dose
  PK plasma parameters
Measure the area under the concentration-time curve from zero up to a definite time t after administration (AUCt) | Pre-dose to 24 hours post-dose
  PK Plasma Parameters

SECONDARY OUTCOMES:
measurement of Pharmacokinetic parameter Area under the curve to infinity after administration (AUCINF) | Pre-dose to 24 hours post-dose
  PK plasma parameters
measurement of Pharmacokinetic parameter time to maximum concentration after administration (tmax) | Pre-dose to 24 hours post-dose
  PK plasma parameters
measurement of Pharmacokinetic parameter of elimination rate after administration (LambdaZ,) | Pre-dose to 24 hours post-dose
  PK plasma parameters
Measurement of Pharmacokinetic parameter elimination of half life after administration ( t1/2Z) | Pre-dose to 24 hours post-dose
  PK plasma parameters
Measurement of heart rate | Pre-dose to 24 hours post-dose
  Vital signs measurements
Measurement of blood pressure | pre-dose to 24 hours post-dose
  vital signs measurement
Measurement of respiration rate | pre-dose to 24 hours post-dose
  vital signs measurement
Measurement of temperature | pre-dose to 24 hours post-dose
  vital signs measurement
Measurement of Saturation Pulse Oxygen (SP02) | pre-dose to 24 hours post-dose
  vital signs measurement

IPD SHARING:
Plan to Share IPD: No